CLINICAL TRIAL: NCT02527811
Title: A Randomized, Controlled Trial Evaluating Efficacy of Perioperative Organ Protection as Well as Safety of Ulinastatin Use in Pediatric Patients Undergoing Open Heart Surgery Through CPB to Treat Complex Congenital Heart Diseases
Brief Title: Ulinastatin Injection in in Pediatric Patients Undergoing Open Heart Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Techpool Bio-Pharma Co., Ltd. (Industry)
Collaborators: Shanghai Children's Medical Center (Other); Guangzhou Women and Children's Medical Center (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Nanjing Children's Hospital (Other); Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GDTP-CDMA-201402
Record Dates: First submitted 2014-12-18; First posted 2015-08-19 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Congenital Heart Diseases
Keywords: ulinastatin; CPB; pediatric
MeSH Terms: conditions — Heart Defects, Congenital | interventions — urinastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ulinastatin group (Experimental): the ulinastatin group will be administered as follows:Ulinastatin 30,000 unit/kg will be diluted into saline solution and administered intravenously in the surgery; Postoperative administration will be 30,000unit/kg divided into 3 regimens until leave ICU.
  Interventions: Drug: Ulinastatin
- control group (No Intervention): patients of control group received conventional therapy,eg,General anesthetic drug and monitoring during the whole process of surgery;Mechanical ventilation and close monitoring to prevent and manage respiratory acidosis and alkalosis and so on.

INTERVENTIONS:
Drug: Ulinastatin — Ulinastatin will be diluted into saline solution and administered intravenously in the intraoperative and postoperative
  Other Names: UTI; urinary trypsin inhibitor; bikunin
  Arms: ulinastatin group

SUMMARY:
1. Explore the efficacy of Ulinastatin use in improving post-operative pulmonary insufficiency and safety in pediatric patients undergoing scheduled CPB open heart surgery to treat Complex Congenital Heart Disease
2. Explore the efficacy of Ulinastatin use in improving intraoperative hemodynamic instability as well as other post-operative organ recuperation and its impact on hospital stay & cost

DETAILED DESCRIPTION:
Pediatric patients diagnosed with Complex Congenital Heart Disease ready to accept scheduled open-heart surgery under cardiopulmonary bypass (CPB).

This study uses randomized (centralized randomization) & controlled design with open label. Eligible subjects will be randomized to receive either study drug (Ulinastatin) or conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with Complex Congenital Heart Disease .
2. Hospitalized children, both gender, aged ≥ 30 days to ≤ 4 years.
3. Preoperative assessment meet with surgical condition.
4. Without signs of Liver, Kidney, and Coagulatory dysfunction.
5. Written informed consent form has been signed by the Legal Guardian.

Exclusion Criteria:

1. Patients will accept minimally invasive surgery or palliative surgery, as well as Major Aortopulmonary Collateral Arteries (MAPCAs);
2. Its decided that subject needs to undergo second surgery in a short period of time, or underwent other major surgery.
3. Subjects with known hypersensitivity to study medication (Ulinastatin for Injection) or patients with highly allergic history.
4. Though meeting the study inclusion criteria, the Legal Guardian reject to sign on informed consent. Or at the discretion of study investigator/coinvestigator that the subjects is not appropriate to be included in the study.

Ages: 30 Days to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Dynamic changes of arterial oxygen tension / inspired oxygen fraction (PaO2/FiO2) ratio | Participants will be followed for the duration of ICU, an expected average of 5 days
  Dynamic changes of PaO2/FiO2 ratio will be observed in every 4 hours interval during post-operative ICU stay period

SECONDARY OUTCOMES:
The time of the PaO2/ FiO2 Ratio ≥300 post surgery | Participants will be followed for the duration of ICU, an expected average of 5 days
The proportion of the PaO2/ FiO2 Ratio ≥300 post surgery | Participants will be followed for the duration of ICU, an expected average of 5 days
Monitoring arterial hydrogen ion concentration | Participants will be followed for the duration of ICU, an expected average of 5 days
Monitoring record of mean blood pressure | Intraoperative and Postoperative,an expected average of 6 days
Monitoring record of central venous pressure | Intraoperative and Postoperative,an expected average of 6 days
Analysis proinflammatory cytokines Interleukin 1 | Preoperative and Postoperative on day1 ,day3 and day5

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, MD, Study Chair — Shanghai Children's Medical Center
Locations (5):
- China (5):
  - General Hospital of Guangzhou Millitary Command, Guangzhou, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Shanghai Children's Medical Center, Shanghai
  - Children's Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided